CLINICAL TRIAL: NCT00669890
Title: Gemtuzumab Ozogamicin in Combination With Busulfan and Cyclophosphamid and Allogenic Stem Cell Transplantation in Patients With High Risk CD33+ Acute Myelogenous Leukemia/Myelodysplastic Syndrome/Juvenile Myelomonocytic Leukemia
Brief Title: Allogenic Stem Cell Transplantation in Patients With High Risk CD33+ AML/MDS/JMML
Acronym: High Risk
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Professor of Pediatrics, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA2533; CHNY-01-515 (Other: CU)
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Acute Myeloid Leukemia; Juvenile Myelomonocytic Leukemia; Myelodysplastic Syndrome
Keywords: AML; JMML; MDS; Allogenic Atem Cell Transplant; Gemtuzumab Ozogamicin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes | interventions — Gemtuzumab; Busulfan; Cyclophosphamide; thymoglobulin; Tacrolimus; Mycophenolic Acid; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study 515 (Experimental)
  Interventions: Drug: Gemtuzumab Ozogamicin; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Thymoglobulin; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Methotrexate

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Dose Escalation
  Other Names: Gemtuzumab
Drug: Busulfan — Conditioning Regimen
  Other Names: Busulfex
Drug: Cyclophosphamide — Conditioning Regimen
  Other Names: Endoxan; Cytoxan
Drug: Thymoglobulin — (Unrelated Donors only)
  Other Names: ATG
Drug: Tacrolimus — GVHD Prophylaxis
  Other Names: FK506
Drug: Mycophenolate Mofetil — GVHD Prophylaxis
  Other Names: MMF
Drug: Methotrexate — GVHD Prophylaxis
  Other Names: MTX

SUMMARY:
The addition of gemtuzumab ozogamicin (GO) in combination with Busulfan/Cyclophosphamide followed by AlloSCT in patients with high risk CD33+ AML/JMML/MDS will be safe and well tolerated.

This study will attempt to determine the maximum tolerated dose of the immune therapy (gemtuzumab) when given in combination with the myeloablative (high dose) drugs used in this study for allogeneic stem cell transplant. (Part A)

DETAILED DESCRIPTION:
Gemtuzumab Ozogamicin (CMA-676) is a chemotherapeutic agent consisting of recombinant humanized anti-CD33 antibody conjugated with calicheamicin, a highly potent cytotoxic antitumor antibiotic. The antibody portion of Gemtuzumab binds specifically to the CD33 antigen, a sialic acid-dependent adhesion protein expressed on the surface of leukemia blasts, normal and leukemic myeloid colony-forming cells, including leukemic clonogenic precursors, but excluding pluripotent hematopoietic stem cells and nonhematopoietic cells. This results in formation of the complex that is internalized, upon which calicheamicin derivative is released with in the lysosomes of the myeloid cell. The free calicheamicin derivative then binds to the DNA, resulting in DNA double strand breaks and consequential cell death.

ELIGIBILITY:
Eligibility

Inclusion Criteria:

Disease Status

* AML Induction Failure
* AML in 1st, 2nd, or 3rd Relapse (>10% bone marrow blasts)
* AML greater than or equal to 3rd CR
* MDS with >6% bone marrow blasts at diagnosis
* Secondary MDS with less than or equal to 5% bone marrow myeloblasts at diagnosis
* JMML with >6% bone marrow myeloblasts at diagnosis

Disease Immunophenotype Patients (AML only) receiving gemtuzumab ozogamicin must express minimum of >10% or =10% CD33 positivity. Patients with <10% CD33 positivity will not receive gemtuzumab ozogamicin.

Organ Function

Patients must have adequate organ function as defined below:

* Adequate renal function defined as:
* Serum creatinine <1.5 x normal, or
* Creatinine clearance or radioisotope GFR 40 ml/min/m2 or >60 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range
* Adequate liver function defined as:
* Total bilirubin 1.5 x normal, or SGOT (AST) or SGPT (ALT) <2.0 x normal or =2.0 x normal
* Adequate cardiac function defined as:
* Shortening fraction of >27% by echocardiogram, or
* Ejection fraction of >47% by radionuclide angiogram or echocardiogram
* Adequate pulmonary function defined as:
* DLCO >55% or =55% by PFT
* For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% on room air

Exclusion Criteria:

* Patients with active CNS AML/JMML/MDS disease at time of conditioning therapy
* Female patients who are pregnant (positive HCG)
* Karnofsky <50% or Lansky <50% if 10 years or less
* Age >65 years
* Has received gemtuzumab in the previous 30 days or has not recovered from prior gemtuzumab therapy.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2004-05; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose or tolerable dose of Gemtuzumab Ozogamicin (anti-CD33 immunotoxin) therapy combined with Busulfan/ Cyclophosphamide in the conditioning regimen prior to AlloSCT in patients with high risk CD33+ AML/JMML/MDS | 1 year

SECONDARY OUTCOMES:
Changes, if applicable, of minimal residual disease (cytogenetics, FISH, RT-PCR) in patients with high risk CD33+ AML/JMML/MDS after AlloSCT. | 1 year
Progression Free Survival (PFS), overall survival (OS), and disease free survival (DFS), (if applicable), following GO, Bu/CY and AlloSCT in patients with high risk CD33+ AML/JMML/MDS. | 1 year
Quality of life before and after GO, Bu/CY conditioning and AlloSCT in patients with high risk CD33+ AML/JMML/MDS | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Study Chair — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital of NYP, New York, New York, United States

REFERENCES:
- See also: (Click on "Morgan Stanley Children's Hospital" and then "Clinical Services" and then "Blood & Marrow Transplantation") — http://www.childrensnyp.org